CLINICAL TRIAL: NCT05879042
Title: Effects of Different Stretching Types on Gastrocnemius Muscle Viscoelastic Properties and Performance
Brief Title: Effects of Stretching Types on Gastrocnemius
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kubra Koce (Other)
Responsible Party: Sponsor-Investigator, Kubra Koce, Lecturer, Istinye University
Organization: Istinye University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 22-143
Record Dates: First submitted 2023-05-18; First posted 2023-05-30 (Actual); Last update posted 2023-08-09 (Actual); Status verified 2023-08

CONDITIONS: Stretch
MeSH Terms: interventions — Muscle Stretching Exercises

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group 1 (Experimental): Static Stretching
  Interventions: Other: Static Stretching
- Group 2 (Experimental): Dynamic Stretching
  Interventions: Other: Dynamic Stretching
- Group 3 (Experimental): PNF Stretching
  Interventions: Other: PNF Stretching
- Group 4 (Sham Comparator): Sham stretching
  Interventions: Other: Sham stretching

INTERVENTIONS:
Other: Static Stretching — Participants will be placed in the maximum dorsiflexion position of the ankle of the dominant side lower extremities. At this last point, it will be held in a static position for 30 seconds. A total of 10 repetitions will be done, with 5-10 seconds rest between repetitions.
  Arms: Group 1
Other: Dynamic Stretching — Participants will be positioned by placing their hands on the edge of the standing wall. They will be asked to try to increase normal ankle motion in a controlled manner using their own body weight. The stretching position will be held for 30 seconds and a total of 10 repetitions will be done. There will be 5-10 seconds rest between repetitions.
  Arms: Group 2
Other: PNF Stretching — For the lateral head of the gastrocnemius muscle, the dominant side lower extremities of the participants will be placed in the extension-adduction-external position. For the medial head of the gastrocnemius muscle, the dominant side lower extremities of the participants will be placed in the extension-abduction-internal rotation position. Participants will be asked to actively go as far as they can in the opposite direction from the starting position (flexion-abduction-internal rotation for the lateral head; flexion-adduction-external rotation for the medial head). When the participant returns to the starting position after reaching the final point, the practitioner will apply the hold-relax technique and will be asked to stay in this position for 10 seconds.
  Arms: Group 3
Other: Sham stretching — Sham stretching will be applied to the calf area. While the participant is lying prone, they will wait 30 seconds in a static position without applying any stretching to the calf area before reaching the end point of the joint range of motion.
  Arms: Group 4

SUMMARY:
Stretching is the process of positioning certain muscles and related soft tissues of the body in a position that will lengthen them. In addition to increasing the range of motion of stretching, different stretching on many functional (maximum isometric torque, muscle-tendon stiffness, passive-resistive torque, viscoelastic deformation) or structural parameters (muscle stiffness, tendon stiffness, muscle fascicle length, pennation angle, neuromuscular relaxation) We can make changes using methods.

Static stretching usually involves actively or passively moving a limb to the full range of motion, holding this stretched position for 15-60 seconds, and then repeating it 2-4 times. Dynamic stretching encompasses all body movements and involves actively moving the active joints through the range of motion in a controlled manner. PNF stretching is known to be more effective than other stretching techniques as it increases both passive and active flexibility and improves joint range of motion in the short term.

The appropriate evaluation of muscle characteristics and keeping a regular record are very important for the course of rehabilitation, clinical decisions, the creation of an appropriate treatment plan, and the evaluation of treatment practices. Objective evaluation methods are needed to measure the functional state of the muscles, that is, their viscoelastic properties. Myotonometric measurement, which is a painless, objective, and non-invasive measurement method, allows the measurement of muscle tone, elasticity, and stiffness. The myotonometer device is a portable handheld device used to measure the stiffness of soft tissues, including muscles and tendons, using a non-invasive approach. It is a device that is easy to use, fast, and very suitable for the purpose. Based on this information, the aim of our study is to evaluate the effects of different stretching types on gastrocnemius muscle viscoelastic properties and performance.

ELIGIBILITY:
Inclusion Criteria:

* Be between the ages of 18-45
* Volunteer to participate in the study

Exclusion Criteria:

* Those who have had major surgery or trauma related to the musculoskeletal system, especially the ankle and calf region
* Those with neurological disease
* Those with rheumatic disease in the active period
* Those with systemic diseases (Diabetes, hypothyroidism, infection, malignancy...)
* Those with serious psychological problems (BDI score of 30 and above)
* Those with contraindications to stretching (acute inflammations, viral and bacterial infections, infectious diseases, fever, deep vein thrombosis, active malignant disease, aneurysms)
* Those who received physiotherapeutic intervention in the ankle and calf region in the last 6 months
* Obesity (BMI≥30 kg/m2)

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2023-05-30 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-08-08 (Actual)

PRIMARY OUTCOMES:
Muscle Tone and Stiffness | 3 weeks
  Muscle tone and stiffness will be evaluated with a myotonometer. The myotonometer was developed for the objective measurement of mechanical muscle properties. Myotonometry reflects the viscoelastic properties of the muscle such as tone and stiffness by creating oscillation in the muscle fiber and is an acceptable and reliable method for measuring the mechanical properties of the muscle in young adults. The device measures muscle tone as the natural oscillation frequency (Hz) calculated as Hz = 1/T; where T is the oscillation time measured in seconds. Muscle stiffness (N/m) is related to the maximum acceleration of oscillation and tissue deformation recorded by the transducer. Myotonometer can measure the firmness of tissues 2 cm below the epidermis.
Forward Jumping Test on One Leg | 3 weeks
  The One Leg Forward Jumping Test will be used to measure the sudden explosive force and performance of the M.Gastrocnemius muscle. Participants will be asked to jump forward as far as possible on one leg. The measurement will be repeated 3 times bilaterally, and the maximum jumping distance will be recorded in cm.

SECONDARY OUTCOMES:
Joint Range of Motion: | 3 weeks
  Ankle dorsiflexion and plantarflexion movements will be measured bilaterally with a digital goniometer. Measurements will be repeated 3 times and the average value will be recorded in degrees.
Isolated Gastrocnemius Shortness Evaluation | 3 weeks
  The gastrocnemius muscle shortness evaluation of the participants will be done bilaterally while in the supine position with the Silfverskiold method and digital goniometer. The knee joint will be positioned in full extension and 90° flexion, the ankle dorsiflexion will be passive while the subtalar joint is in the neutral position, and the fixed arm of the universal goniometer will be measured on the fibula shaft and the movable arm will be positioned on the fifth metatarsal shaft. The resulting angles will be recorded and evaluated in degrees.

CONTACTS AND LOCATIONS:
Locations (1):
- Istinye University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No